CLINICAL TRIAL: NCT07089927
Title: AVATARS: Adolescent and Young Adult Virtual Art Therapy Assisted Re-Integration During Cancer Survivorship
Brief Title: Virtual Art Therapy Assisted Re-Integration to Improve Biopsychosocial Outcomes in Adolescent and Young Adult Cancer Survivors, AVATARS Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AVATARS; NCI-2025-04978 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-012402 (Other: Mayo Clinic Institutional Review Board); AVATARS (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Neoplasm; Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Art Therapy; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (Virtual art therapy) (Experimental): Patients complete virtual art therapy sessions, over 60 minutes, every 1-2 weeks, for 4 sessions. Patients then receive a 3D printed replica of their avatar.
  Interventions: Procedure: Art Therapy; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Procedure: Art Therapy — Complete virtual art therapy sessions. When complete the participant will receive a 3D printed replica of the avatar.
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests the feasibility, usability and acceptability of a virtual art therapy assisted re-integration (AVATARS) intervention to improve biopsychosocial outcomes, such as anxiety, depression, resilience, emotional regulation, stress, and cognition, among adolescent and young adult (AYA) cancer survivors. AYA cancer survivors (especially those treated at adult cancer centers) historically experience worse psychosocial outcomes and lack age appropriate psychosocial support compared to older adult cancer survivors. Creative art therapy accesses the limbic system to provide a corrective emotional experience in response to trauma and can help patients visually express depression, anxiety, and existential fears, process traumatic events, and regain agency and control. The AVATARS intervention may be a feasible, useable and acceptable way to improve biopsychosocial outcomes among AYA cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate the AVATARS intervention's feasibility, usability, and acceptability among a sample of AYA cancer survivors.

II. Investigate the preliminary efficacy of the AVATARS intervention on biopsychosocial outcomes (i.e. anxiety, depression, resilience, emotional regulation, stress, and cognition) in AYA cancer survivors.

OUTLINE:

Patients complete virtual art therapy sessions, over 60 minutes, every 1-2 weeks, for 4 sessions. Patients then receive a 3D printed replica of their avatar.

After completion of study treatment, patients are followed up at 1 and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-25 years of age at the time of enrollment and able to provide informed consent
* Mild or greater depression [Patient Health Questionnaire (PHQ-A) score > 5]
* Received a cancer diagnosis during the past year, or completed cancer treatment within the past five years (extended survivorship)
* Have access to an electronic device which supports Zoom videoconferencing (e.g., personal device or public library access)
* Able to read and write in English

Exclusion Criteria:

* Participation in art therapy within the past 12 months
* Visual or cognitive impairment which may impede completing the art project or the data collection measures
* Endorsed suicidality (via PHQ-A or otherwise)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility-Enrollment | Up to 4 months
  Assessed via the percentage of eligible participants who enroll in this study.
Feasibility-Completion | Up to 4 months
  Assessed via the percentage of participants who complete at least 75% of the intervention sessions.
Intervention Usability Scale | Up to 4 months
  Assessed by the Intervention Usability Scale. It is a 10-item questionnaire with questions answered on a 5-point scale where 1 = strongly disagree and 5 = strongly agree. Higher scores indicate greater usability.
Acceptability-Exit Interview | Up to 6 months
  Participants will be invited to provide feedback about their experience during brief (e.g., 20- 30 minute) scripted open-ended question exit interviews. Participants perspectives about the intervention, administration format, and schedule will be used to refine the intervention.
Change in Anxiety | T1 (at baseline within 48 hours of recruitment), T2 (within 72 hours post session two, and T3 (within 72 hours post session four), T4 (1 month post session four), and an optional measement at T5 (2 months post session four
  Assessed via State-Trait Anxiety Inventory. This is a 20-item questionnaire related to the current anxiety. Questions are answered on a scale of 1 to 4 where 1 = none at all, 2= a little, 3 = somewhat and 4 = very much so. Higher scores indicate greater feelings of anxiety.
Change in Depression | T1 (at baseline within 48 hours of recruitment), T2 (within 72 hours post session two, and T3 (within 72 hours post session four), T4 (1 month post session four), and an optional measement at T5 (2 months post session four
  Assessed via Patient Health Questionnaire for Adolescents (PHG-A). This is a 13-item questionnaire related to feelings of depression. Questions 1-9 relate to the last two weeks and are answered on a scale of 0 to 3 where 0=Not at all, 1=Several days, 2=More than half of the days and 3=Nearly every day. Lower scores indicate lesser feelings of depression. Two questions relate to feelings of depression over the past year, and two questions relate to suicidal thoughts.
Change in Resilience | T1 (at baseline within 48 hours of recruitment), T2 (within 72 hours post session two, and T3 (within 72 hours post session four), T4 (1 month post session four), and an optional measement at T5 (2 months post session four
  Assessed via Connor Davidson Resilience Scale 10 (CD-RISC-10), a 10-item questionnaire related to resilience over the past month. Questions are answered on a scale of 0 to 4, where 0=not true at all, 1=rarely true, 2=sometimes true, 3=often true and 4=true nearly all the time. Higher scores indicate greater resilience.
Change in Emotional regulation | T1 (at baseline within 48 hours of recruitment), T2 (within 72 hours post session two, and T3 (within 72 hours post session four), T4 (1 month post session four), and an optional measement at T5 (2 months post session four
  Assessed via Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire related to difficulties in emotional regulation. Questions area answered on a 5-point scale (almost never to almost always). A higher score indicates greater difficulties in emotional regulation.

CONTACTS AND LOCATIONS:
Overall Officials: C. Robert Bennett, PhD, RN, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota